CLINICAL TRIAL: NCT06159777
Title: Pre- and Post-operative Compared to Post-operative Only Polyethylene Glycol 3350 for Minimally Invasive Urogynecologic Surgery
Brief Title: Pre-operative Polyethylene Glycol 3350 for Minimally Invasive Urogynecologic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, David Sheyn, Associate professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20231417
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Constipation; Surgical Procedure, Unspecified; Prolapse; Female
Keywords: postoperative constipation; minimally invasive surgery; apical prolapse; prolapse
MeSH Terms: conditions — Constipation; Prolapse | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-operative (Experimental): Participants will be instructed to take 17 grams of powder Polyethylene glycol 3350 (PEG) every day starting 3 days prior to scheduled surgery date and continue to take 17 grams of PEG every day for 7 days following the day of surgery. Participants will be allowed to titrate up or down the amount of PEG used as needed and instructed to record all doses of PEG used.
  Interventions: Drug: Polyethylene Glycol 3350
- Post-operative (Active Comparator): Participants will be instructed to take 17 grams of powder PEG* every day for 7 days starting the day of surgery. Participants will be allowed to titrate up or down the amount of PEG used as needed and instructed to record all doses of PEG used.
  Interventions: Drug: Polyethylene Glycol 3350

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — *Polyethylene glycol 3350 (PEG) will be used within it's FDA indication and dosing for constipation. Each 17-gram dose of PEG is to be mixed in 8oz of liquid.
  Other Names: Miralax

SUMMARY:
The goal of this clinical trial is to test the use of a laxative before surgery in women having surgery to fix pelvic prolapse that do not have constipation.

The main question it aims to answer is: Does use of a laxative before surgery lessen the discomfort of bowel movements after surgery? Participants will be asked to complete questionnaires before and after surgery. Researchers will compare using the laxative before and after surgery versus only after surgery to see if there is less discomfort with bowel movements after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if there is a difference in bother related to constipation between a pre-operative versus post-operative start of a bowel regimen for patients undergoing surgery for pelvic organ prolapse This will be a multi-institution, single-blind, randomized control trial utilizing questionnaires and chart review to evaluate effect of pre-operative bowel regimen on post-operative constipation.

1. Study team and surgeons will be blinded to group assignments, participants will not be.
2. Participants will be randomized after consent is obtained, and at least 1 week prior to planned surgery, via computer-generated blocks in a 1:1 ratio between study group (pre-operative and post-operative use) and control group (post-operative only use) of polyethylene glycol 3350 (PEG)

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned female sex at birth undergoing an apical prolapse procedure including: sacrocolpopexy, sacrospinous ligament suspension, uterosacral ligament suspension, or colpocleisis. Planned urogynecologic procedure may include hysterectomy, adnexectomy, colporrhaphy, perineorrhaphy, or treatment of stress urinary incontinence.
* Planning to undergo primary procedure as above via minimally invasive route: vaginal or laparoscopic (including robotic-assisted). Including those that have an unplanned conversion intraoperatively of minimally invasive route to open laparotomy.

Exclusion Criteria:

* Diagnosis of irritable bowel syndrome, inflammatory bowel disease, slow transit constipation, obstructed defecation, or symptomatic constipation at time of study screening and recruitment. (Slow transit constipation and obstructed defecation defined as per American Gastroenterological Association 2013 constipation statement. Symptomatic constipation defined as any of the following: Bristol Stool Scale score of 1 or 2, PAC-SYM score greater than 1.0, self-reported 2 or less bowel movements per week.)
* Current use of pharmacologic laxative agent ≥1x/week (prescription or OTC) for the treatment of constipation symptoms
* Allergy or intolerance to polyethylene glycol 3350
* Planning to undergo surgery via laparotomy
* Scheduled for any concurrent non-urogynecologic procedure, ex abdominoplasty
* History of large bowel resection, surgical treatment of constipation, or anal sphincter surgery
* History of sacral neuromodulation
* Current or prior radiation therapy to the abdomen or pelvis
* Current or prior diagnosis of malignancy
* Unable to provide informed consent

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
PAC-SYM | Pre-operative, 1 week post-operative, 2 weeks post-operative
  Patient assessment of constipation symptoms (PAC-SYM) is a validated 12-item questionnaire with reported average score 0-4.

SECONDARY OUTCOMES:
PAC-QOL: Patient assessment of constipation quality of life measure | Pre-operative, 2 weeks post-operative
Time to first bowel movement | 1 week post-operative
  after surgery in approximate hours/days
Doses of PEG used | 1 week post-operative, 2 weeks post-operative
  polyethylene glycol 3350 (PEG) doses of 17 grams powder mixed in 8oz of liquid
Rescue laxative use | 1 week post-operative, 2 weeks post-operative
  Use of additional laxatives or enemas
Satisfaction with pain after surgery | 1 week post-operative
  Satisfaction with pain after surgery

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No